CLINICAL TRIAL: NCT03120546
Title: A Randomized Comparison of Cervical Spine Motion During Tracheal Intubation Using Video Laryngoscope or Rigid Video Stylet in Patients With Simulated Cervical Immobilization
Brief Title: Cervical Spine Motion During Tracheal Intubation: Video Laryngoscope vs Rigid Video Stylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: McGrath vs Optiscope
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Intubation
Keywords: cervical spine motion; video laryngoscope; rigid video stylet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): rigid video stylet intubation - video laryngoscope intubation
  Interventions: Device: rigid video stylet intubation; Device: video laryngoscope intubation
- Group B (Experimental): video laryngoscope intubation - rigid video stylet intubation
  Interventions: Device: rigid video stylet intubation; Device: video laryngoscope intubation

INTERVENTIONS:
Device: rigid video stylet intubation — intubation using rigid video stylet
Device: video laryngoscope intubation — intubation using video laryngoscope

SUMMARY:
In this study, investigators are going to compare cervical spine motion during tracheal intubation using video laryngoscope or rigid video stylet in patients with simulated cervical immobilization.

DETAILED DESCRIPTION:
In patients with an unstable cervical spine, neck extension during tracheal intubation may result in harmful events such as spinal cord injury. Thus, it is important to minimize cervical spine motion in these patients. In this randomized crossover study, investigators are going to compare cervical spine motion during tracheal intubation using video laryngoscope or rigid video stylet in patients with simulated cervical immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years undergoing elective endovascular cerebral aneurysm coiling to general anesthesia in a neuroangiography suite

Exclusion Criteria:

* Patients with upper airway abnormalities such as inflammation, abscesses, tumors, polyps, and trauma
* Patients with a medical history of gastroesophageal reflux disease and previous airway surgery, at high risk for aspiration, coagulation disorders, or a Hunt Hess grade of 3-5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
maximum cervical spine motion | during tracheal intubation
  maximum angles measured at the occiput-C1, C1-C2, C2-C5 segments

SECONDARY OUTCOMES:
intubation time | during tracheal intubation
  time interval between insertion of the device into the oral cavity and its removal
number of intubation trial | during tracheal intubation
  number of intubation trial

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, M.D., Ph. D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No